CLINICAL TRIAL: NCT02127697
Title: A Randomized, Double-blind, Parallel Group, 52-week Study Evaluating the Efficacy, Safety and Tolerability of NVA237 in Patients With Poorly Controlled Asthma
Brief Title: Study of Efficacy and Safety of NVA237 in Patients With Poorly Controlled Asthma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNVA237B2301
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Asthma
Keywords: Asthma, poorly controlled asthma, LAMA, Long-Acting Muscarinic Antagonist, Glycopyrronium, Glycopyrronium bromide, Anticholinergic
MeSH Terms: conditions — Asthma | interventions — Glycopyrrolate; Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NVA237 (Experimental): Participants will receive NVA237 once daily in addition to their background therapy during the 52- week treatment period. All participants will receive salbutamol/ albuterol as rescue medication.
  Interventions: Drug: NVA237; Drug: salbutamol/ albuterol
- Placebo (Placebo Comparator): Participants will receive placebo to NVA237 in addition to their background therapy during the 52-week treatment period. All participants will receive salbutamol/ albuterol as rescue medication.
  Interventions: Drug: Placebo to NVA237; Drug: salbutamol/ albuterol

INTERVENTIONS:
Drug: NVA237 — NVA237 capsules for inhalation, delivered via Concept1 once daily
  Arms: NVA237
Drug: Placebo to NVA237 — Placebo to NVA237 delivered via Concept1 once daily
  Arms: Placebo
Drug: salbutamol/ albuterol — Taken as rescue medication

SUMMARY:
The study will assess efficacy, safety and tolerability of NVA237 compared to placebo in patients with poorly controlled asthma over 52 weeks of treatment.

DETAILED DESCRIPTION:
The study will assess efficacy and safety of NVA237 compared to placebo, in addition to background therapy with LABA/ICS in patients with poorly controlled asthma.

ELIGIBILITY:
Inclusion Criteria:

Written informed consent must be obtained before any assessment is performed; Male and female adult patients aged 18 to <75 years; Patients with a diagnosis of asthma (according to GINA 2012) for a period of at least 5 years prior screening; The diagnosis of asthma must have been made before the patient was 40; Increase in forced expiratory volume in 1 second (FEV1) of ≥ 12% and ≥ 200 mLs within 30 minutes after administration of 400 µg salbutamol/360 µg albuterol (or equivalent dose); Pre-bronchodilator FEV1 of ≥ 50 and ≤ 80% of the predicted normal value for the patient; Patients who qualify for treatment (according to GINA 2012) and have been treated with a stable dose of a fixed dose inhaled corticosteriod (ICS) and long-acting β2 agonist (LABA) combination for at least 4 weeks prior to screening. Patient must be using a total daily dose of ICS of ≥800 μg/day of budesonide of equivalent; All patients must be symptomatic with a mean ACQ-5 score ≥ 1.5 at Visit 101 and Visit 102; A documented history of one or more asthma exacerbations in the previous 12 months that required either treatment with additional or increased dose of systemic corticosteroids for at least 3 days, or an emergency room visit, or hospital treatment, or intubation

Exclusion Criteria:

Contraindicated for treatment with, or having a history of reactions/ hypersensitivity to any of the following inhaled drugs, drugs of a similar class, or any component thereof:

Muscarinic antagonist agents, sympathomimetic amines, lactose or any of the other excipients of the study drug, long and short acting beta-2 agonists, corticosteroids; Women of child-bearing potential; Resting QTcF ≥ 450 ms (male) or ≥ 460 ms (female) at Visit 101 (assessed by central reader) and at Visit 102 (assessed by investigator at the site); Patients with a body mass index (BMI) of more than 40 kg/m2; Patients who have clinically significant renal, cardiovascular (such as but not limited to unstable ischemic heart disease, NYHA Class III/IV left ventricular failure, myocardial infarction, arrhythmia, neurological, endocrine, immunological, psychiatric, gastrointestinal, hepatic, or hematological abnormalities which could interfere with the assessment of the efficacy and safety of the study treatment; Patients with narrow-angle glaucoma, symptomatic benign prostatic hyperplasia or bladder-neck obstruction or moderate to severe renal impairment or urinary retention (BPH patients who are stable on treatment can be considered); Patients who have had an asthma exacerbation that required either treatment with additional or increased dose of systemic corticosteroids for at least 3 days, or an emergency room visit, or hospital treatment, or intubation in the 6 weeks prior to screening; Patients who have smoked or inhaled tobacco products within the 6 month period prior to screening, or who have a smoking history of greater than 10 pack years (Note:10 pack years = 1 pack /day x 10 yrs., or ½ pack/day x 20 yrs.); Patients with a history of chronic lung diseases other than asthma, including (but not limited to) chronic obstructive pulmonary disease, bronchiectasis, sarcoidosis, interstitial lung disease, cystic fibrosis, and tuberculosis (unless tuberculosis is confirmed as no longer active by imaging); Patients on Maintenance Immunotherapy (desensitization) for allergies must have been so for at least 3 months prior to run-in, and must be expected to remain unchanged throughout the course of the study;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Trough Forced Expiratory Volume in 1 Second (FEV1) at Week 26 | Week 26
  Spirometry testing will be performed in accordance with American Thoracic Society standards. Trough FEV1 defined as the mean of two measurements at 23 hours 15 minutes and 23 hour 45 minutes post dosing.

SECONDARY OUTCOMES:
Time to First Moderate or Severe Asthma Exacerbation Over 52 Weeks of Treatment | 52 weeks
  Asthma exacerbations are considered to be moderate if treatment with rescue systemic corticosteroids for greater than or equal to 3 days as outpatient or less than or equal to 24 hour emergency room visit was required. Asthma exacerbations are considered severe if treatment with rescue systemic corticosteroids for greater than or equal to 3 days and hospitalization or emergency department visit greater than 24 hours were required or death due to asthma. The time to the first moderate or severe asthma exacerbation is the study day on which the patient experienced first moderate or severe asthma exacerbation.
Asthma Control Questionnaire (ACQ-7) Overall Score at Week 26 | Week 26
  Asthma symptoms will be evaluated by the Asthma Control Questionnaire (ACQ-7). The ACQ has six questions to be answered by the patient, each with a 7 point scale (0-good control, 6-poor control), and one item where the actual pre-bronchodilator FEV1 value expressed in % of predicted FEV1. The overall score is an average of the 7 items.
Quality of Life as Assessed by Standardised Asthma Quality of Life Questionnaire (AQLQ(S)) Over 52-Week Treatment Period. | Week 12, Week 26, Week 52
  There are 32 questions in the AQLQ and they are in 4 domains (symptoms, activity limitation, emotional function and environmental exposure). Each question will be answered on a 7 point scale (1-totally limited/problems all the time, 7-not at all limited/no problems). The overall AQLQ score is the mean of all 32 responses, and the individual domain scores are the means of the items in those domains (a minimum domain / overall score of 1 = Severely impaired whereas a maximum domain / overall score of 7 = not impaired at all). A positive change from baseline score indicates improvement.
Quality of Life Assessment With St. George's Respiratory Questionnaire (SGRQ) Over 52-Week Treatment Period | Week 12, Week 26, Week 52
  SGRQ is a health related quality of life questionnaire consisting of 50 items in three components: symptoms, activity, and impacts. The lowest possible value is zero and the highest 100. Higher values correspond to greater impairment in quality of life.
Shortened Version of the Asthma Control Questionnaire (ACQ-6) | Week 4, Week 8, Week 12, Week 26, Week 39, Week 52
  This shortened version of the asthma control questionnaire (symptoms plus β2-agonist) consists of 6 items (nighttime waking, symptoms on waking, activity limitation, shortness of breath, wheeze and rescue short-acting β2-agonist use) between 0 and 6 (0 = maximum control; 6 = no control ) and a total score is the mean of 6 items.
Shortened Version of the Asthma Control Questionnaire (ACQ-5) | Week 4, Week 8, Week 12, Week 26, Week 39, Week 52
  This shortened version of the asthma control questionnaire (symptoms only) consists of 5 items (nighttime waking, symptoms on waking, activity limitation, shortness of breath, and wheeze) between 0 and 6 (0 = maximum control; 6 = no control) and a total score is the mean of 5 items.
Peak Forced Expiratory Volume in 1 Second (FEV1) Over 52 Weeks of Treatment | Day 1, Week 4, Week 26, Week 52
  Spirometry will be conducted according to internationally accepted standards. Peak FEV1= the maximum FEV1 recorded in the period between 0 minutes and 3 hours post dose.
Forced Expiratory Volume in 1 Second (FEV1) Standardized (With Respect to Length of Time) Area Under the Curve (AUC0-3h) Over 52 Weeks of Treatment | Day 1, Week 4, Week 26, Week 52
  FEV1 will be measured with spirometry conducted according to internationally accepted standards. Measurements will be made at 5, 15, and 30 minutes; and 1, 2, and 3 hours post-dose.
Predose Forced Expiratory Volume in 1 Second (FEV1) Over 52 Weeks of Treatment | Week 2, Week 4, Week 8, Week 26, Week 39, Week 52
  FEV1 will be measured with spirometry conducted according to internationally accepted standards. Predose FEV1 defined as the mean of FEV1 at -45 minutes and -15 minutes before the morning dose.
Trough Forced Expiratory Volume in 1 Second (FEV1) Over 52 Weeks of Treatment | Day 2, Week 4, Week 26, Week 52
  FEV1 will be measured with spirometry conducted according to internationally accepted standards. Trough FEV1 defined as the mean of FEV1 23 hours 15 minutes and the 23 hours 45 minutes post dose.
Mean Daily Number of Puffs of Rescue Medication Over 52 Weeks of Treatment | 52 Weeks
  Participants will maintain a diary to record the number of puffs of rescue Short-acting B2 agonist (SABA) used in the previous 24 hours to treat asthma symptoms.
Rate of Moderate or Severe Asthma Exacerbation | 52 Weeks
  Rate of moderate or severe exacerbations per year = total number of moderate or severe exacerbations / total number of treatment years
Rate of Severe Asthma Exacerbation | 52 Weeks
  Rate of severe exacerbations per year = total number of moderate or severe exacerbations / total number of treatment years
Time To First Severe Asthma Exacerbation | 52 Weeks
  Asthma exacerbations are considered to be severe if treatment with rescue systemic corticosteroids for greater than or equal to 3 days and hospitalization or emergency department visit greater than 24 hours required or death due to asthma. The time to the first severe asthma exacerbation = the study day on which the patient experienced first severe asthma exacerbation.
Time To First Asthma Exacerbation (Mild, Moderate, or Severe) | 52 Weeks
  Asthma exacerbation are considered Mild if treatment with inhaled or nebulized Short-acting B2 agonist (SABA), increase in inhaled corticosteroid only, or requires less than 3 days of systemic corticosteroids. Asthma exacerbations are considered to be moderate if treatment with rescue systemic corticosteroids for greater than or equal to 3 days as outpatient or less than or equal to 24 hour emergency room visit required. Asthma exacerbations are considered severe if treatment with rescue systemic corticosteroids for greater than or equal to 3 days and hospitalization or emergency department visit greater than 24 hours required or death due to asthma. The time to the first mild, moderate, or severe asthma exacerbation = the study day on which the patient experienced first asthma exacerbation of any severity.
Rate of Asthma Exacerbation (Mild, Moderate, or Severe) | 52 Weeks
  Rate of mild, moderate or severe exacerbations per year = total number of moderate or severe exacerbations / total number of treatment years
Morning Daily Peak Expiratory Flow (PEF) Over 52 Weeks of Treatment | Every 3 Months, 52 Weeks
  Peak Expiratory Flow (PEF) will be measured every morning within 15 minutes of waking and before dosing using a peak flow meter, and recorded in the patient diary.
Evening Daily Peak Expiratory Flow (PEF) Over 52 Weeks of Treatment | Every 3 Months, 52 Weeks
  Peak Expiratory Flow (PEF) will be measured every evening using a peak flow meter, and recorded in the patient diary.
Asthma Control Diary (ACD) Symptom Score Over 52-Week Treatment Period | Every 3 Months, 52 Weeks
  The mean symptom score for ACD is defined as the sum of daily symptom scores divided by number of days where diary records were made. The daily symptom score for ACD is defined as the mean of the responses to the 5 symptom questions for any day with ACD questions answered.
Lung Function Assessed by Forced Expiratory Volume for 1 Second (FEV1) | Week 1, Week 2, Week 4, Week 8, Week 12, Week 26, Week 39, Week 52
  FEV1 will be measured with spirometry conducted according to internationally accepted standards.
Forced Vital Capacity (FVC) | Week 2, Week 4, Week 8, Week 12, Week 26, Week 39, Week 52
  Forced Vital Capacity (FVC) is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. FVC will be assessed via spirometry. A positive change from baseline in FVC indicates improvement in lung function.
Asthma Control Questionnaire (ACQ-7) Over 52 Weeks of Treatment | Week 4, Week 8, Week 12, Week 26, Week 39, Week 52
  Asthma symptoms will be evaluated by the Asthma Control Questionnaire (ACQ). The ACQ has six questions to be answered by the patient, each with a 7 point scale (0-good control, 6-poor control), and one item where the actual pre-bronchodilator FEV1 value expressed in % of predicted FEV1. The overall score is an average of the 7 items.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals